

# STATISTICAL ANALYSIS PLAN

| Title | Phase 3b Open-label Extension Study to Evaluate the Safety<br>and Efficacy of Aceneuramic Acid Extended-Release<br>(Ace-ER) Tablets in Patients with GNE Myopathy (GNEM)<br>or Hereditary Inclusion Body Myopathy (HIBM) |
|---|---|
| Protocol: | UX001-CL302 |
| <b>Protocol Version:</b> | Amendment 1 (17 June 2016) |
| <b>Investigational Product:</b> | Aceneuramic Acid Extended-Release (Ace-ER) Tablets |
| Phase: | 3b |
| Sponsor: | Ultragenyx Pharmaceutical Inc. |
| | 60 Leveroni Court |
| | Novato, CA, USA 94949 |
| Author: | PPD |
| | <b>Biostatistics Consultant</b> |

15 June 2017

Version 1.0

Date:

**Version Number:** 



# TABLE OF CONTENTS

| AI | BBRE | EVIATIONS | 5 |
|---|---|---|---|
| 1 | INTRODUCTION | | |
| 2 | STU | JDY OBJECTIVE(S) | 8 |
| | 2.1 | Overall Safety Objective(s) | 8 |
| | 2.2 | Overall Efficacy Objective(s) | 8 |
| 3 | STU | JDY DESIGN | 9 |
| | 3.1 | Study Population | 10 |
| | 3.2 | Dosage and Administration | 10 |
| | 3.3 | Blinding and Randomization Methods | 10 |
| | 3.4 | Stratification Factors | 10 |
| | 3.5 | Sample Size Considerations | 10 |
| | 3.6 | Interim Analysis | 10 |
| | 3.7 | Data Monitoring Committee | 10 |
| 4 | STU | JDY ENDPOINTS AND COVARIATES | 11 |
| | 4.1 | Safety Endpoints | 11 |
| | | 4.1.1 Primary Safety Endpoint | 11 |
| | | 4.1.2 Other Safety Endpoints | 11 |
| | 4.2 | Efficacy Endpoints | 11 |
| 5 | DEF | FINITIONS | 14 |
| | 5.1 | Baseline | 14 |
| | 5.2 | Subgroup | 14 |
| 6 | ANA | ALYSIS SETS | 15 |
| 7 | DA | ΓA SCREENING AND ACCEPTANCE | 16 |
| | 7.1 | General Principles | 16 |
| | 7.2 | Handling of Missing and Incomplete Data | 16 |
| | | 7.2.1 Missing Date of the Last Dose of Investigational Product | 16 |



| | | 7.2.2 | Missing Efficacy Data | 16 |
|---|---|---|---|---|
| | | 7.2.3 | Missing Dates Information for Adverse Events and Concomitant<br>Medications | 16 |
| | | 7.2.4 | Missing Causal Relationship to Investigational Product for Adverse Events | 17 |
| | | 7.2.5 | Visit Time Windows | 17 |
| | 7.3 | Handli | ng of Multiple Measurements in HHD | 17 |
| | 7.4 | Testing | g/Validation Plan | 17 |
| | 7.5 | Softwa | re | 17 |
| 8 | STA | TISTIC | AL METHODS OF ANALYSES | 18 |
| | 8.1 | Genera | ıl Principles | 18 |
| | 8.2 | Subjec | t Disposition | 19 |
| | 8.3 | Protoco | ol Deviations | 19 |
| | 8.4 | Demog | graphic and Baseline Characteristics | 20 |
| | 8.5 | Investi | gational Product Administration | 20 |
| | | 8.5.1 | Extent of Exposure | 20 |
| | | 8.5.2 | Measurement of Treatment Compliance | 20 |
| | 8.6 | Efficac | y Analysis | 20 |
| | 8.7 | Safety | Analysis | 21 |
| | | 8.7.1 | Adverse Events | 21 |
| | | | 8.7.1.1 Adverse Events to Monitor | 22 |
| | | 8.7.2 | Concomitant Medication | 22 |
| | | 8.7.3 | Clinical Laboratory Parameters | 22 |
| | | 8.7.4 | Vital Signs | 22 |
| | | 8.7.5 | Physical and Neurological Exams | 22 |
| | | 8.7.6 | Interval History | 23 |
| | | 8.7.7 | Suicidal Ideation | 23 |
| | | 8.7.8 | Pregnancy Test | 23 |



| 9 | REFERENCES | 24 |
|---|---|---|
| 10 | APPENDICES | 25 |
| | 10.1 Summary of Efficacy Endpoints and Analyses | 25 |
| | 10.2 Missing Observation in Hand Held Dynamometry and GNEM-FAS | 28 |
| | 10.3 Computation Formula for Derived HHD Variables | 31 |
| | 10.3.1 Predicted Normal HHD Muscle Strength | 32 |
| | 10.4 Summary of Efficacy Assessment in Parent Studies and in Current Study CL302 | 37 |
| | 10.5 Schedule of Events | 39 |
| | 10.6 Adverse Events to Monitor | 42 |
| | 10.6.1 Gastrointestinal MedDRA Query | 42 |
| | 10.6.2 Liver-Related Investigations | 43 |
| | 10.7 Table templates for efficacy and safety analysis presentation | 44 |
| Lis | et of Tables | |
| Tal | ble 4.2.1: Efficacy Assessments Performed by Parent Study | 13 |
| Tal | ble 8.1.1: Analysis Presentation | 19 |
| Lis | st of Figures | |
| Fig | gure 3.1: Study Schema | 9 |



#### **ABBREVIATIONS**

6MWT Six Minute Walk Test

Ace-ER Aceneuramic Acid Extended-Release

AE adverse event

ATC Anatomical Therapeutic Chemical

CK creatine kinase

C-SSRS Columbia-Suicide Severity Rating Scale

CTCAE Common Terminology Criteria for Adverse Events

DMC data monitoring committee

DMRV distal myopathy with rimmed vacuoles

ET early termination

GEE generalized estimating equation

GNE/MNK glucosamine (UDP-N-acetyl)-2-epimerase/N-acetylmannosamine

kinase

GNEM GNE Myopathy

GNEM-FAS GNE Myopathy Functional Activities Scale

HHD hand held dynamometry

HIBM hereditary inclusion body myopathy

INQoL Individualized Neuromuscular Quality of Life Questionnaire

IP investigational product

LEC lower extremity composite

ManNAc N-acetyl-D-mannosamine

MedDRA Medical Dictionary for Regulatory Activities

MCS mental component summary

CTCAE Common Terminology Criteria for Adverse Events

PCS physical component summary

PT preferred term

qHS at the time of sleep (i.e., at bedtime)

SA sialic acid

SAE serious adverse event

SAP Statistical Analysis Plan



SAS Statistical Analysis System

SD standard deviation

SF-36v2 Short Formc-36 Health Survey version 2

SOC system organ Class

TEAE treatment-emergent adverse event

TID three times per day

UEC upper extremity composite

US United States



#### 1 INTRODUCTION

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within the UX001-CL302 original protocol dated 10 February 2016 and the UX001-CL302 Protocol Amendment 1 dated 17 June 2016. Should there be a difference between the SAP and the protocol with respect to analysis methods, the SAP will take precedence over the protocol.



# 2 STUDY OBJECTIVE(S)

The study objective is to evaluate the long-term safety and efficacy of Ace-ER treatment of GNE Myopathy subjects.

# 2.1 Overall Safety Objective(s)

Primary objective is to evaluate the long-term safety of 6 g/day Ace-ER treatment in subjects with GNE Myopathy.

# 2.2 Overall Efficacy Objective(s)

Secondary objective is to evaluate the long-term effect of 6 g/day Ace-ER treatment in subjects with GNE Myopathy.



#### 3 STUDY DESIGN

This open-label extension study of will assess the long-term safety and efficacy of Ace-ER treatment over a period of 24 months. Approximately 180 subjects from the UX001-CL202, UX001-CL301, and UX001-CL203 studies will be eligible to enroll in the study.

Subjects will take 4 tablets (500 mg Ace-ER each for 2 g per dose) orally 3 times per day (TID). The dose should be taken with food (i.e. within 30 minutes after a meal or snack). Subjects being treated with 12 g/day Ace-ER in UX001-CL202 will be transitioned to 6 g/day Ace-ER dose in this protocol. Treatment will be administered for a total of 24 months. Study visits will occur every 8 weeks for 24 weeks and then every 6 months for subjects enrolling from UX001-CL202 or UX001-CL301. For subjects enrolling from UX001-CL203 studies, study visits will occur every 6 months. The schedule of assessments is shown in Appendix 10.4.

Safety will be evaluated by review of the incidence and frequency of AEs and SAEs and clinically significant changes in interval history, physical examination results, vital signs, clinical laboratory test results, the Columbia Suicide Severity Rating Scale (C-SSRS) (Posner et al. 2011), and concomitant medications.

Blood samples will be collected to evaluate biomarkers (for example sialylation of serum proteins before and after treatment) to determine their utility in predicting clinical outcomes.

Efficacy will be evaluated based on assessments used in the parent study from which subjects roll over (subjects enrolling from UX001-CL202 will follow the same schedule of events as subjects who roll over from UX001-CL301), and include dynamometry as a measure of muscle strength and patient- and clinician-reported outcome measures as indicators of physical functioning and quality of life. For UX001-CL202 subjects, assessments that cannot be safely performed by a subject due to disease progression should not be administered.

A study schema demonstrating the enrolling patient populations and scheduled study visits is shown in Figure 3.1.

Adult GNEM
patients who
complete
UX001-CL202,
UX001-CL301, or
UX001-CL203
studies

Ace-ER 6 g/day
N= ~165

M2<sup>a</sup> M4<sup>a</sup> M6 M12 M18 M24

\*Only for subjects who roll-over from UX001-CL202 or UX001-CL301

Figure 3.1: Study Schema



# 3.1 Study Population

This study will be conducted in adults who have previously documented mutations in the gene for the GNE/MNK enzyme leading to a diagnosis of GNEM (variously termed HIBM, DMRV, or Nonaka disease). These patients have an impaired ability to synthesize endogenous SA, which leads to muscle weakness and atrophy. Consequently, this is the relevant population for testing SA replacement therapy, and for determining if SA replacement leads to improved protein and lipid sialylation and stabilized or improved muscle structure and performance.

Individuals who have ingested N-acetyl-D-mannosamine (ManNAc) or similar other SA-producing compounds during the 60 days prior to the Screening Visit will be excluded as it could confound interpretation of the results.

#### 3.2 Dosage and Administration

Each Ace-ER tablet contains 500 mg of SA in an extended release formulation for a total weight of 1200 mg/tablet. The drug will be administered by the oral route and will be divided into a TID regimen: 4 tablets taken in the morning, early evening, and before bedtime (qHS). The dose should be taken with food (i.e., within 30 minutes after a meal or snack).

Treatment will be administered for a total of 24 months (96 weeks).

# 3.3 Blinding and Randomization Methods

This is open-label extension study consists of one treatment arm. All subjects will be treated with Ace-ER 6 g/day. Randomization and blinding are not applicable.

#### 3.4 Stratification Factors

No stratification factors are planned.

#### 3.5 Sample Size Considerations

The current study is primarily designed to evaluate safety and the sample size is intended to provide the maximum amount of information regarding UX001 tolerability along with indicators of long-term safety and efficacy in this patient population. Approximately 180 adult subjects with GNEM are expected to roll-over from UX001-CL202, UX001-CL301, and UX001-CL203 studies to participate in this extension study.

#### 3.6 Interim Analysis

No interim analysis is planned for this study.

#### 3.7 Data Monitoring Committee

No formal DMC is planned for this study in the protocol. Conduct of the study and safety of the patients will be monitored by Ultragenyx on a regular basis.



#### 4 STUDY ENDPOINTS AND COVARIATES

All data are collected according to the schedule of assessments (Appendix 10.4).

Overall safety endpoints serve to evaluate the long-term safety of 6 g/day Ace-ER treatment in subjects with GNE Myopathy (primary objective).

Overall efficacy endpoints serve to evaluate the long-term effect of 6 g/day of Ace-ER treatment in subjects with GNEM.

# 4.1 Safety Endpoints

# 4.1.1 Primary Safety Endpoint

The primary endpoint of the study is the incidence and frequency of AEs and SAEs assessed as related to Ace-ER over the duration of the study.

# 4.1.2 Other Safety Endpoints

Other safety endpoints include clinically significant changes from baseline to scheduled time points in the following:

- Interval History
- Vital signs
- Physical examination results
- Clinical laboratory results
- C-SSRS (a measure of suicidal ideation and behavior)
- Concomitant medications

Drug concentration endpoints will be evaluated for the following:

- Changes from baseline in free SA level in serum;
- Changes from baseline in urine SA level;
- Frequency and percentage of subjects with the presence of ManNac detected from urine testing.

#### 4.2 Efficacy Endpoints

Efficacy evaluations will be based on the parent study (UX001-CL202, UX001-CL301, or UX001-CL203) from which the subjects enroll. Subjects enrolling from UX001-CL202 follow the same schedule of visits for the efficacy assessments as subjects who roll over from UX001-CL301. Subjects enrolling from UX001-CL203 follow a different schedule of visits.



# For subjects enrolling from UX001-CL202 and UX001-CL301:

#### Primary Clinical Efficacy Endpoint:

• Changes from baseline in upper extremity composite score (UEC) based on bilateral strength recorded in the following muscle groups: gross grip, shoulder abductors, elbow flexors, and elbow extensors as measured by dynamometry. The UEC is derived from the sum of the average of the right and left total force values (measured in kg);

# **Secondary Clinical Efficacy Endpoints:**

- Changes from baseline in the scores on the mobility domain of GNEM-FAS;
- Change from baseline in the scores on the upper extremity domain of GNEM-FAS;
- Changes from baseline in lower extremity composite score (LEC) based on bilateral strength recorded in the following muscle groups: knee flexors, hip flexors, hip extensors, hip abductors and hip adductors as measured by dynamometry. The LEC is derived from the sum of the average of the right and left total force values;
- Change from baseline in the number of stands in the Sit-to-Stand test;
- Changes from baseline in the number of lifts in 30 second weighted arm lift;
- Changes from baseline in meters walked in 6MWT and percent predicted distance based on normative data for age and gender;
- Changes from baseline in total force and percent predicted total force in the Knee Extensors. The percent predicted total force value will be determined based on reference equations adjusting for age, gender, height, and weight.

#### **Tertiary Efficacy Endpoints:**

- Changes from baseline in UEC and LEC percent predicted based on reference equations adjusting for age, gender, height, and weight;
- Changes from baseline in bilateral total force and percent predicted total force for each individual muscle group included in the UEC and LEC;
- Changes from baseline in the score on self-care domain on GNEM-FAS;
- Changes from baseline in the total score on GNEM-FAS;
- Change from baseline in in the total score from a 45-item self-report questionnaire (INQoL) on the impact of key muscle disease symptoms on the ability to perform basic activities of daily living, functional independence, relationships and overall well-being;
- Changes from baseline in CK levels in serum to assess the degree of reduction of CK levels observed as a surrogate for muscle injury.



# For subjects enrolling from UX001-CL203:

#### Primary Clinical Efficacy Endpoints:

- Changes from baseline in the mobility domain of GNEM-FAS Expanded Version;
- Changes from baseline in the upper extremity domain of GNEM-FAS Expanded Version;
- Changes from baseline in the self-care domain of GNEM-FAS Expanded Version;
- Changes from baseline in the total scores of GNEM-FAS Expanded Version;
- Changes from baseline in upper extremity muscle strength and percent predicted in the following muscle groups: grip, key pinch, shoulder abductors and wrist extensors as measured by HHD
- Changes from baseline in lower extremity muscle strength and percent predicted in the knee extensors as measured by HHD

#### **Exploratory endpoints:**

- Changes from baseline in 8 subscales and summary scores (PCS and MCS) in health-related quality of life as assessed by using Short Form Health Survey – 36 (SF-36v2);
- Changes from baseline in creatine kinase (CK) and serum aceneuramic acid.

Assessments, upon which efficacy endpoints are based on, are shown in Table 4.2.1. Detailed information on efficacy endpoints and visit schedules by study can be found in Appendix 10.1.

Table 4.2.1: Efficacy Assessments Performed by Parent Study

| | CL202 and CL301 | CL203 |
|---|---|---|
| Assessment | Week 0, 8, 16, 24, 48, 72, 96 | Week 0, 24, 48, 72, 96 |
| Functional | HHD* 6MWT Sit-to-Stand Test Weighted Arm Lift Test GNEM FAS | HHD^ GNEM FAS expanded version |
| QoL Questionnaire | INQoL | SF-36 short form |
| Biomarker | CK Free serum SA Urine ManNAc | |

<sup>\*</sup> Measured by HHD, the Upper Extremity Composite (UEC) Score is based on gross grip, shoulder abductors, elbow flexors, and elbow extensors. The Lower Extremity Composite (LEC) Score is based on knee flexors, hip flexors, hip abductors, and hip adductors.

<sup>^</sup> Measured by HHD, UEC is not defined in this study for analysis, since different muscle groups from the other two studies are measured. Lower extremity muscle strength of knee extensors is included.



#### 5 DEFINITIONS

#### 5.1 Baseline

Two baselines are defined for the statistical analysis variable derivations.

- Current study baseline is defined as the last observed value before the first dosing of the study drug for CL302.
- Parent study baseline is defined as the last observed value before the first dosing of the IP study drug from CL202, CL203, or CL301 depending on which study the subject was enrolled from.

Current study baseline is defined for all safety summaries and analyses.

Efficacy summaries and analyses will be performed upon the parent study baseline and the current study baseline as specified in Table 8.1.1.

#### 5.2 Subgroup

The following subgroups are defined for this study:

- Gender (Male and Female)
- Age (above and below median)
- Ethnicity (small groups may be combined)
- Genetic Mutation
  - Genotype: Homozygote, Heterozygote, and Compound Heterozygote
  - Mutation type: Exon and Intron

Genetic mutation subgroup analysis will be done for the following primary efficacy endpoints: the changes from baseline in UEC score in subjects enrolled from CL301 and CL202; and the changes from baseline in lower extremity muscle strength of knee extensors in subjects enrolled from CL203.

Gender, age, and ethnicity subgroup summaries will be done to support the safety.



#### **6 ANALYSIS SETS**

Three analysis sets are defined for the study.

**Full Analysis Set**: The full analysis set will include all subjects with a CL302 baseline measurement and at least one post-baseline measurement in CL302. This set will be used for the efficacy analysis.

**Safety Analysis Set**: The safety analysis set consists of all subjects who receive at least one dose of study drug in CL302. This set will be used for safety analysis.

**Sialic Acid Analysis Set**: The SA analysis set will consist of all subjects with evaluable free serum SA levels in CL302.



#### 7 DATA SCREENING AND ACCEPTANCE

# 7.1 General Principles

Data will be reviewed periodically. And any questionable data will be reported to the clinical data manager promptly for query and resolution.

#### 7.2 Handling of Missing and Incomplete Data

Missing clinical outcome data can occur for multiple reasons, including missed subject visits and scales or measures with missing item scores. Missing and incomplete data will be identified through the data quality review plan for this study. Missing and incomplete data will be identified for investigation, and possible resolution, by Data Management prior to the study database lock or snapshot. Unless specified otherwise, only the observed data (not imputed data) will be presented in listings.

#### 7.2.1 Missing Date of the Last Dose of Investigational Product

When the date of the last dose of investigational product is found missing for a subject, all efforts should be made to obtain the date from the Investigator. If after all efforts are made it is still missing, the last dosing visit date will be used as the last dose date.

# 7.2.2 Missing Efficacy Data

Details of missing HHD observations for individual muscle groups and individual questions for GNEM-FAS are provided in Appendix 10.2.

# 7.2.3 Missing Dates Information for Adverse Events and Concomitant Medications

The following conventions will be used to impute missing portions of dates for adverse events and concomitant medications. Note that the imputed values outlined here may not always provide the most conservative date. In those circumstances, the imputed value may be replaced by a date that will lead to a more conservative analysis.

#### Missing Start Dates

- If the day is unknown, then:
  - o If the month and year match the first dose of investigational product start date month and year in this study, then impute the day of the first dose date.
  - Otherwise, assign the first day of the month.
- If the month is unknown, then:
  - o If the year matches the year of the first dose of investigational product date in this study, then impute the month and day of the first dose date in this study.
  - o Otherwise, assign 'January'



• If the year is unknown, then the date will not be imputed and will be assigned a missing value.

If the imputed date is earlier than birth date, then birth date will be used

#### Missing Stop Dates

- If the day is unknown, then assign the last day of the month.
- If the month is unknown, then assign 'December.'
- If the year is unknown, then the date will not be imputed and will be assigned a missing value.

If the resulting end date is after the date of study completion / discontinuation/ data cutoff, set the imputed end date as the date of study completion / discontinuation/ data cutoff.

# 7.2.4 Missing Causal Relationship to Investigational Product for Adverse Events

If the causal relationship to the investigational product is missing for an AE that started on or after the date of the first dose of investigational product, a causality of "definitely related" will be assigned. The imputed values for causal relationship to investigational product will be used for the incidence summary; the values will be shown as missing in the data listings.

#### 7.2.5 Visit Time Windows

There is no visit time window applied to handle the missing values for a scheduled visit. Nominal visits will be used for by-visit analyses. If an unscheduled visit has to be used, the principle of proximity will be applied.

#### 7.3 Handling of Multiple Measurements in HHD

Each muscle strength is assessed three times in Hand Held Dynamometry (HHD) measurement. The highest value of the three will be used for summary and derivation of efficacy endpoints.

#### 7.4 Testing/Validation Plan

Data will be reviewed by cross functional team periodically and issues will be addressed by clinical data management.

#### 7.5 Software

SAS<sup>®</sup> software version 9.2 or higher will be used to perform statistical analyses unless otherwise specified.



#### 8 STATISTICAL METHODS OF ANALYSES

# 8.1 General Principles

All statistical tests will be two-sided and a difference resulting in a p-value of less than or equal to 0.05 will be considered statistically significant. All p-values will be rounded to and displayed in four decimals. If a p-value less than 0.0001 occurs, it will be shown in the table as <0.0001.

Continuous variables will be summarized by number of subjects and mean, SD/SE, median, minimum, and maximum values. Categorical variables will be summarized by number and percentage. No imputation on missing data will be made, unless stated otherwise.

Data collected will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included in the data listings.

Post-hoc exploratory analyses not identified in this SAP may be performed to further examine the study data. These analyses will be clearly identified as such in the final clinical study report. The SAP will not be amended for post-hoc or additional analyses identified after planned analyses are completed. Similarly, additional tables and figures may be defined to further evaluate study results and the SAP will not be amended to list them.

Efficacy analyses will be presented by the parent study as illustrated in Table 8.1.1: UX001-CL301, CL202 or CL203. Different efficacy endpoints at different scheduled time points were collected depending on which parent study the subjects were enrolled from.

Safety analyses will be presented by the parent studies and overall as illustrated in Table 8.1.1. Subjects enrolling from UX001-CL301 will be further examined by the treatment group assigned in the parent study: placebo, Ace-ER 6 g/day, and All.

Table 8.1.1 also provides the guidance for the treatment groups to be displayed for biomarker analyses as well as efficacy analyses and safety analyses, which have been described above. Baseline used for the analyses are specified as well. Example table templates are provided in Appendix 10.6 for efficacy and safety.



**Table 8.1.1: Analysis Presentation** 

| Analysis Category | Analysis Set | Parent Study | Treatment Group | Baseline Applied |
|---|---|---|---|---|
| | | CL301 | Placebo* | |
| | | | Ace-ER 6 g/day | Parent Study Baseline |
| | | | Placebo* | |
| Week 96/ET efficacy | | | ACE-ER 6 g/day | Current Study |
| analysis | Full Analysis Set | | All | Baseline |
| Week 96/ET efficacy analysis | Full Analysis Set | CL202 | Ace-ER 6 g/day | Current Study<br>Baseline |
| | | CL203 | Ace-ER 6 g/day | Parent Study Baseline |
| Week 96 /ET efficacy analysis | Full Analysis Set | | Ace-ER 6 g/day | Current Study<br>Baseline |
| | | CL301 | Placebo* | |
| | | | Ace-ER 6 g/day | |
| | | | All | |
| | | CL202 | | |
| Week 96/ET safety | Safety Analysis | CL203 | | Current Study |
| analysis | Set | Total | Ace-ER 6 g/day | Baseline |
| | | CL301 | | |
| | | CL202 | | |
| Week 96/ET analysis | Sialic Acid | CL203 | | Current Study |
| on biomarkers | Analysis Set | Total | Ace-ER 6 g/day | Baseline |

<sup>\*</sup> This refers to the enrolled subjects who had received placebo treatment in parent study CL301.

#### 8.2 Subject Disposition

All subjects screened for the study will be used for reporting of disposition. Subject disposition summaries will include the number and percentage of subjects who are included in the safety, efficacy, and SA analysis sets; the number and percentage of subjects who received study drug treatment, completed the study or discontinued the study (with reasons) will be summarized by parent study and total.

#### **8.3** Protocol Deviations

Major protocol deviations will be summarized. All protocol deviations will be listed.



# 8.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized descriptively for the full analysis set.

- Gender
- Age
- Age at start of parent study
- Race
- Ethnicity
- Height (cm)
- Weight (kg)
- Genotype: Homozygote, Heterozygote, and Compound Heterozygote
- Mutation type: Exon and Intron

# 8.5 Investigational Product Administration

# 8.5.1 Extent of Exposure

The total number of doses administered, the total dose administered, and the total treatment duration will be summarized for the Safety Analysis Set. The calculation will be based on the current study baseline unless otherwise specified.

Study medication dispensing and treatment compliance will also be listed.

# **8.5.2** Measurement of Treatment Compliance

Dosing compliance for a CL302 study period is defined as:

Actual total dosage taken during CL302 / Planned dosage for CL302 \* 100%.

Descriptive statistics will be reported for compliance on the Safety Analysis Set.

#### 8.6 Efficacy Analysis

Efficacy analyses will use generalized estimating equation (GEE) (Hanley et al. 2003) to evaluate trends over time with respect to the changes from baseline for all continuous efficacy endpoints. Baseline will be included as a covariate in the model. GEE will be the primary analysis method for all repeated measures endpoints. The statistical analyses will be reported in summary tables, figures, and data listings. Statistical tests will be 2-sided at the alpha=0.05 significance level.



Efficacy analysis will be based on the full analysis set.

Additional efficacy analyses may be performed for subjects enrolled in CL301 by incorporating data from both the parent study and the current study to compare the placebo versus UX001 treatment groups using the methodology described in (Hu et al. 2007). Such analyses examine the extended treatment effect of UX001 on the placebo subjects who now are taking UX001 in the extension study.

Parent study baseline will be used to evaluate the long-term study drug effect from the parent study drug administration, except for subjects enrolling from CL202.

Current study baseline will be used to evaluate the continuous long-term study drug effect going on after the parent study.

# 8.7 Safety Analysis

The safety analysis will be performed on the safety analysis set. Descriptive statistics will be provided for safety reporting by parent study and overall.

#### 8.7.1 Adverse Events

All AEs recorded from the time the subject signs the informed consent through the safety follow-up will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 17.1 or beyond).

The following AEs were collected:

- All AEs;
- All SAEs;
- Treatment-related AEs;
- Treatment-related SAEs:
- AEs leading to the discontinuation of study drug or discontinuation of study;
- Deaths.

The number and proportion of subjects with any treatment-emergent adverse events (TEAEs) (defined generally as any AE started on or after the first dose of study drug) will be summarized by System Organ Class (SOC), Preferred Term (PT), severity, grade, outcome and relationship to treatment for the following types of AEs. Additional summaries of subject incidence (by preferred term) will also be provided.

An AE continued from the parent study would be excluded since they were summarized in the parent study. However, if an AE continued from the parent study and the severity changed to worse will be considered as a TEAE and be summarized.



The severity of AEs will be based on Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03. If an AE cannot be graded based on CTCAE, the investigator will assign a severity based on 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = Death.

For those AEs that occurred more than once during the study, the maximum severity or highest grade will be used to summarize the subject incidence.

Detailed listings for all AEs, serious AEs, AEs leading to the discontinuation of study, and death will also be provided.

Subgroup analyses by gender, age (above and below median), and ethnicity (small group may be combined) will be performed to support the safety in GNEM patients.

#### **8.7.1.1** Adverse Events to Monitor

Adverse events to be monitored are included in Appendix 10.5 by MedDRA preferred terms in categories of gastrointestinal AEs and liver-related investigations.

Tables summarizing patient incidents for the monitored adverse events will be generated.

#### 8.7.2 Concomitant Medication

The number and percent of concomitant medications in CL302 will be summarized by ATC class and preferred term (per WHO-drug dictionary) in the safety analysis set.

If a subject took a specific medication multiple times or took multiple medications within a specific therapeutic class, that subject will be counted only once for the coded drug name or therapeutic class.

#### 8.7.3 Clinical Laboratory Parameters

Descriptive statistics for clinical laboratory values and changes from the CL302 baseline values at each visit will be presented. The number and percentage of abnormalities for each lab parameter at each assessment time point will be reported.

#### 8.7.4 Vital Signs

Descriptive statistics for vital signs including blood pressures, respiration rate, and heart rate and changes from CL302 baseline values at each scheduled visit and at the end of study will be presented. All results of vital signs will be listed.

#### 8.7.5 Physical and Neurological Exams

A complete physical examination including neurological exam is performed at CL302 baseline. At post-baseline visit, a subset of physical examination (brief exam including



general appearance, cardiovascular exam, and respiratory exam) is conducted. The number and percentage of abnormal findings will be summarized for the complete physical exam. The number and percentage of deficit findings will be summarized for the neurological exam. The number and percentage of abnormal findings for the brief exam will be summarized for post-baseline visits in a similar fashion.

# 8.7.6 Interval History

The Interval history in CL302 will be summarized for number and percentage of patients who reported changes at each visit from the last visit.

#### 8.7.7 Suicidal Ideation

The Columbia Suicide Severity Rating Scale (C-SSRS) is a standardized rating instrument used to assess the suicidal ideation and behavior in an at-risk population and will be administered at each visit. Any 'Yes' response from C-SSRS will be listed.

#### 8.7.8 Pregnancy Test

Pregnancy test will be conducted at the scheduled study visit and the results will be provided in a listing.



#### 9 REFERENCES

Bohannon, RW. 1997a. "Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants." *Age Ageing* 26 (1):15-9.

Bohannon, RW. 1997b. "Reference values for extremity muscle strength obtained by handheld dynamometry from adults aged 20 to 79 years." *Arch.Phys.Med.Rehabil.* 78 (1):26-32.

Hanley, JA, Negassa, A, Edwardes, MD, and Forrester, JE. 2003. "Statistical analysis of correlated data using generalized estimating equations: an orientation." *Am J Epidemiol* 157 (4):364-75.

Hu, Z, and Follmann, D. 2007. "Statistical methods for active extension trials." *Stat Med* 26 (12):2433-48.

NIMS. 1996. "Muscular weakness assessment: use of normal isometric strength data. The National Isometric Muscle Strength (NIMS) Database Consortium." *Arch Phys Med Rehabil* 77 (12):1251-5.

Peters, MJ, van Nes, SI, Vanhoutte, EK, Bakkers, M, van Doorn, PA, Merkies, IS, Faber, CG, and PeriNom, SSg. 2011. "Revised normative values for grip strength with the Jamar dynamometer." *J Peripher Nerv Syst* 16 (1):47-50.

Posner, K, Brown, GK, Stanley, B, Brent, DA, Yershova, KV, Oquendo, MA, Currier, GW, Melvin, GA, Greenhill, L, Shen, S, and Mann, JJ. 2011. "The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults." *Am J Psychiatry* 168 (12):1266-77.

Stoll, T, Huber, E, Seifert, B, Michel, BA, and Stucki, G. 2000. "Maximal isometric muscle strength: normative values and gender-specific relation to age." *Clin Rheumatol* 19 (2):105-13.

Visser, J, Mans, E, de Visser, M, van den Berg-Vos, RM, Franssen, H, de Jong, JM, van den Berg, LH, Wokke, JH, and de Haan, RJ. 2003. "Comparison of maximal voluntary isometric contraction and hand-held dynamometry in measuring muscle strength of patients with progressive lower motor neuron syndrome." *Neuromuscul Disord* 13 (9):744-50.



# 10 APPENDICES

# 10.1 Summary of Efficacy Endpoints and Analyses

| Test / Instrument Endpoint | | Type of analysis | Time points for<br>Assessment | Statistical<br>approach at<br>week 96/ET<br>analysis |
|---|---|---|---|---|
| Subjects enrolling | Subjects enrolling from UX001-202 and UX001-301 | | | |
| Physical therapy –<br>Hand-held<br>Dynamometry<br>(HHD) | The changes from baseline in Upper Extremity Composite (UEC) Score based on bilateral strength recorded in the following muscle groups: gross grip, shoulder abductors, elbow flexors, and elbow extensors | Primary analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |
| GNEM Functional Activities Scale (GNEM-FAS) | Changes from baseline on Upper Extremity Domain score Changes on Mobility Domain score | Secondary<br>efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |
| Physical therapy –<br>Hand-held<br>Dynamometry<br>(HHD) | Changes from baseline in lower extremity composite score (LEC) based on bilateral strength recorded in the following muscle groups: knee flexors, hip flexors, hip extensors, hip abductors and hip adductors. Changes from baseline in total force and percent predicted total force in the Knee Extensors. | Secondary<br>efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |
| Sit to Stand | Change from baseline in the number of stands in the Sit-to-Stand test | Secondary efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |
| Weighed Arm<br>Lift Test | Changes from baseline in the number of lifts in 30 second weighted arm lift tests | Secondary<br>efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |
| 6-Minute Walk<br>Test | Changes from baseline in meters walked in 6MWT and percent predicted | Secondary<br>efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | GEE Model |



| Test /<br>Instrument | Endnoint | | Time points for<br>Assessment | Statistical<br>approach at<br>week 96/ET<br>analysis |
|---|---|---|---|---|
| Physical therapy –<br>Hand-held | Changes from baseline in UEC and LEC percent predicted based on reference equations adjusting for age, gender, height, and weight. | Tertiary efficacy | Weeks 8, 16, 24, | Summary statistics |
| Dynamometry<br>(HHD) | Changes from baseline in bilateral total force and percent predicted total force for each individual muscle group included in the UEC and LEC. | analysis 48, 72, and 96 | Summary statistics | |
| GNEM | Changes from baseline on the total score on the GNEM-FAS | T | W 1 0 16 24 | C |
| Functional<br>Activities Scale<br>(GNEM-FAS) | Changes from baseline on the<br>Self-Care Domain Score on the<br>GNEM-FAS | Tertiary efficacy analysis | Weeks 8, 16, 24, 48, 72, and 96 | Summary statistics |
| Individual Neuromuscular Quality of Life Questionnaire (INQoL) (Not including CL202 subjects) | Changes from baseline on the total score on a 45-item self-report questionnaire on the impact of key muscle disease symptoms on the ability to perform basic activities of daily living, functional independence, relationships and overall well-being | Tertiary efficacy<br>analysis | Weeks 8, 16, 24, 48, 72, and 96 | Summary<br>statistics |
| Creatine Kinase<br>(CK) | Changes from baseline in CK levels in serum to assess the degree of reduction of CK levels observed as a surrogate for muscle injury | Tertiary efficacy<br>analysis | Weeks 8, 16, 24, 48, 72, and 96 | Summary<br>statistics |
| Subjects enrolling from UX001-203 | | | | |
| GNEM Functional Activities Scale (GNEM-FAS) Expanded Version | Changes from baseline in the total scores Changes from baseline in the mobility domain Changes from baseline in the upper extremity domain Changes from baseline in the self-care domain | Primary efficacy<br>analysis | Weeks 24, 48, 72, and 96 | GEE Model |



| Test /<br>Instrument | Endpoint | Type of analysis | Time points for<br>Assessment | Statistical<br>approach at<br>week 96/ET<br>analysis |
|---|---|---|---|---|
| Physical therapy –<br>Hand-held<br>Dynamometry<br>(HHD) | Hand-held Dynamometry Shoulder abductors and wrist extensors | | Weeks 24, 48, 72, and 96 | GEE Model |
| Short Form<br>Health Survey –<br>36 (SF-36v2) | Changes from baseline in 8 subscales and summary scores (PCS and MCS) in SF-36v2 | Exploratory efficacy analysis | Weeks 24, 48, 72, and 96 | Summary statistics |
| Biomarker | Changes from baseline in serum<br>biomarkers: creatine kinase (CK),<br>serum aceneuramic acid | Exploratory efficacy analysis | Weeks 24, 48, 72, and 96 | Summary statistics |



# 10.2 Missing Observation in Hand Held Dynamometry and GNEM-FAS

Imputation rules outlined in this section for dynamometry are defined below and are based on the distinct pattern of muscle weakness associated with GNE Myopathy and the features of the dynamometers used in this study. The most common cause of missing data is muscle weakness severe enough to prevent the subject from registering the minimum amount of force against the dynamometer required to obtain a measurement during a maximum voluntary isometric contraction maneuver. In those cases, the value is imputed to 0, and preserves the ability to calculate the UEC and LEC scores. There are some scenarios in which non-random missing HHD data values result in missing UEC and LEC values. When strength in a particular muscle group exceeds the resistance that can be applied by the administrator, a reliable value cannot be obtained from the dynamometer. This is a recognized limitation of a hand-held device (Visser et al. 2003). In GNE Myopathy, the only muscle group at risk for this scenario is the knee extensors, due to the relative sparing of the quadriceps. All other non-random missing HHD data are related to the clinical condition of the subject at the time of the testing where a test may not be administered due to pain, injury, contracture or another extenuating circumstance that could cause discomfort to the subject. The proposed plan for the handling of this data is intended to provide the most accurate estimate of muscle strength and physical function possible based on knowledge of the disease and the outcome measures obtained during the conduct of previous studies.

Missing observations in HHD for individual muscle group will be imputed based on reason for missing and if the muscle strength measurement is missing on both sides or one side. The table below provides a summary of the imputation rule followed by detailed descriptions.

| Instrument | Missing Reason | Imputation |
|---|---|---|
| HHD missing BOTH sides | Too Weak | 0 |
| | Too Strong | NA, UE/LE composite not computed |
| | Pain | NA, UE/LE composite not computed |
| | Injury | NA, UE/LE composite not computed |
| | Contracture | NA, UE/LE composite not computed |
| | Other | NA, UE/LE composite not computed |
| HHD missing ONE side | Too Weak | 0 |
| | All other reasons | The value from the other side that was measured |



 $Missing\ Reason = Weakness$ 

A value of 0 should be imputed for a W.

- If both sides are W, a value of 0 is assigned to each side and the muscle group IS counted as part of the UE or LE composite.
- If one side is W, a value of 0 is assigned to that side and the 0 is averaged with the value from the other side. The muscle group IS counted as part of the UE of LE composite.

Missing Reason = Contracture

A value of 0 should NOT be imputed for a C. A C is missing data because the test was not performed due to the contracture.

- If both sides are C (which would be rare), then the data for this muscle group is missing and the UE or LE composite will be set to missing.
- If one side is C, then the data is missing from this side and the value from the other side should be used to reflect the total strength for this muscle group. The muscle group IS counted as part of the UE or LE composite.

Missing Reason = Pain

A value of 0 should NOT be imputed for a P. A P is missing data because the test was not performed due to pain.

- If both sides are P, then the data for this muscle group is missing and the UE or LE composite will be set to missing.
- If one side is P, then the data is missing from this side and the value from the other side should be used to reflect the total strength for this muscle group. The muscle group IS counted as part of the UE or LE composite.

Missing Reason = Injury

A value of 0 should NOT be imputed for an I. An I is missing data because the test was not performed due to pain.

- If both sides are I, then the data for this muscle group is missing and the UE or LE composite will be set to missing.
- If one side is I, then the data is missing from this side and the value from the other side should be used to reflect the total strength for this muscle group. The muscle group IS counted as part of the UE or LE composite.

Missing Reason = Too Strong

An S indicates that the test was attempted but that the subject overpowered the administrator and a valid value could not be obtained.



- If both sides are S, then the data for this muscle group is missing and the UE or LE composite will be set to missing.
- If one side is S, then the data is missing from this side and the value from the other side should be used to reflect the total strength for this muscle group. The muscle group IS counted as part of the UE or LE composite.

 $Missing\ Reason = OTHER$ 

No value should be imputed if there is an O.

- If both sides are O, then the data for this muscle group is missing and the UE or LE composite will be set to missing.
- If one side is O, then the data is missing from this side and the value from the other side should be used to reflect the total strength for this muscle group. The muscle group IS counted as part of the UE or LE composite.

When an individual question is missing in GNEM-FAS. The average score is calculated for the domain and then multiplied by the number of questions in the domain:

Mobility Subscale Score = 10 x Sum(Available Items) / Number of Available Items

Upper Extremity Subscale Score = 8 x Sum(Available Items) / Number of Available Items

Self-Care Subscale Score =  $7 \times \text{Sum}(\text{Available Items}) / \text{Number of Available Items}$ 

If a domain has more than 50% (inclusive) items missing ( $\geq$ 5 for Mobility,  $\geq$ 4 for Upper Extremity,  $\geq$ 3 for Self-Care), the domain score will not be calculated. The Total FAS core will only be calculated if all three domain scores are available.



# 10.3 Computation Formula for Derived HHD Variables

**Individual Muscle Strength Average Score** = (left-side measurement + right-side measurement) / 2

**UE Composite Score** = sum( Individual Muscle Strength Average Score for muscle group gross grip, shoulder abductors, elbow flexors and elbow extensors)

**LE Composite Score** = sum(Individual Muscle Strength Average Score for muscle group knee flexors, hip flexors, hip extensors, hip abductors and hip adductors)

**Predicted Normal for Individual Muscle Strength Average Score** = (left-side predicted normal + right-side predicted normal) / 2

**Predicted Normal for UE Composite Score** = sum(Predicted Normal for Individual Muscle Strength Average Score for muscle group gross grip, shoulder abductors, elbow flexors and elbow extensors)

**Predicted Normal for LE Composite Score** = sum(Predicted Normal for Individual Muscle Strength Average Score for muscle group hip flexors, hip extensors, hip adductors and knee flexors)

% of predicted normal HHD values = (Observed strength value/ Predicted normal strength value) \*100%.

Predicted normal HHD values can be derived using the regression equations outlined in Appendix 10.3.1.



# 10.3.1 Predicted Normal HHD Muscle Strength

# **Muscle Strength**

Note: Many of the HHD derived variables detailed below rely on regression equations that have predictor variables in units different than what is found in the analysis datasets. Care will be taken to convert dataset variables to the correct units before they are entered into the prediction equation. The resulting predicted value will then, in turn, be converted to the appropriate unit for analysis.

#### **Hand-Held Dynamometry**

# Shoulder abduction and hip abduction

Regression Equations and Multiple Correlations of Sex, Age, and Weight with Muscle Strength

| Muscle Action | Side | Equation* | R | R <sup>2</sup> |
|---|---|---|---|---|
| Shoulder Abduction | Nondominant | 165.16 – 74.9S – .910A + .126W | .843 | .710 |
| | Dominant | 178.90 – 77.1S – 1.128A + .134W | .843 | .710 |
| Hip Abduction | Nondominant | 203.32 - 73.3S - 1.247A + .192W | .794 | .630 |
| | Dominant | 195.24 - 62.4S - 1.184A + .198W | .764 | .584 |

<sup>(</sup>Bohannon 1997b)

**Note:** Age and weight values collected at the Baseline visit will be used for the calculation of predicted values for shoulder abduction and hip abduction for all study time points.

#### Hip adduction

| Muscle Action | Gender | Side | Age (years) | Equation |
|---------------|--------|-------|----------------|-------------------------|
| Hip Adduction | Female | Left | ≤ 55 | 19.1 – 0.30*(age -55) |
| | Female | Right | <u>≤</u> 55 | 19.5 – 0.00*(age -55) |
| | Female | Left | > 55 | 19.1 – 0.212*(age -55) |
| | Female | Right | > 55 | 19.5 – 0.245*(age - 55) |
| Hip Adduction | Male | Left | <u>&lt;</u> 49 | 31.8 + 0.044*(age – 49) |
| | Male | Right | <u>&lt;</u> 49 | 31.6 - 0.082*(age – 49) |
| | Male | Left | > 49 | 31.8 - 0.280*(age – 49) |
| | Male | Right | > 49 | 31.6 - 0.206*(age – 49) |

(Stoll et al. 2000)

Median strength results in kiloponds (kp) also known as kilogram-force (kgf)

<sup>\*</sup>Muscle strength results in Newtons (N). S, sex (male=0, female=1); A, age (years); W, weight (Newtons).



**Note:** The age category that applies for a subject at the Baseline visit will be used for the calculation of hip adduction predicted values for all study time points.

# Elbow flexion, elbow extension, hip flexion, hip extension, knee flexion, knee extension Regression Equations for Strength Prediction

#### **Muscle Action** Equation - (age \* 0.13) + (gender \* 11.24) + ((weight/height<sup>2</sup>) \* 0.07) + 22.78 Right Elbow Flexion $-(age * 0.11) + (gender * 10.63) + ((weight/height^2) * 0.05) + 19.66$ Left Elbow Flexion $- (age * 0.08) + (gender * 8.33) + ((weight/height^2) * 0.16) + 12.37$ Right Elbow Extension $-(age * 0.07) + (gender * 8.18) + ((weight/height^2) * 0.17) + 11.32$ Left Elbow Extension - (age \* 0.33) + (gender \* 19.19) + ((weight/height<sup>2</sup>) \* 0.66) + 34.44Right Hip Flexion Left Hip Flexion $-(age * 0.29) + (gender * 18.75) + ((weight/height^2) * 0.47) + 36.05$ -(age \* $0.21 + (gender * 15.19) + ((weight/height^2) * 0.14) + 33.52$ Right Hip Extension -(age \* 0.23) + (gender \* 15.02) + ((weight/height<sup>2</sup>) \* 0.17) + 33.88 Left Hip Extension -(age \* 0.16) + (gender \* 8.78) + ((weight/height<sup>2</sup>) \* 0.08) + 22.47 Right Knee Flexion Left Knee Flexion -(age \* 0.17) + (gender \* 7.67) + ((weight/height<sup>2</sup>) \* 0.14) + 21.10 $-(age * 0.38) + (gender * 18.44) + ((weight/height^2) * 0.62) + 34.41$ Right Knee Extension - (age \* 0.38) + (gender \* 17.68) + ((weight/height<sup>2</sup>) \* 0.62) + 33.61 Left Knee Extension

#### (NIMS 1996)

Strength prediction results in kilograms (kg)

Age = years; gender: male = 1, female = 0; weight = kg;; height = meters

**Note:** Age, height and weight values collected at the Baseline visit will be used for the calculation of predicted values for elbow flexion, elbow extension, hip flexion, hip extension, knee flexion and knee extension for all study time points.



# **Gross Grip**

# Normative grip strength values for the Jamar dynamometer for clinical use (in pounds)

| | | Females (n = 35 | 55) | Males (n = 365) | | |
|---|---|---|---|---|---|---|
| Age<br>(years) | Number<br>of<br>subjects | 5 <sup>th</sup> %ile<br>Jamar values<br>(lbs) | Median<br>Jamar values<br>(lbs) | Number of subjects | 5 <sup>th</sup> %ile<br>Jamar values<br>(lbs) | Median<br>Jamar values<br>(lbs) |
| 20 - 29 | 51 | 50 | 62 | 50 | 81 | 100 |
| 30 – 39 | 50 | 49 | 64 | 51 | 80 | 105 |
| 40 – 49 | 50 | 48 | 63 | 50 | 78 | 107 |
| 50 – 59 | 51 | 45 | 61 | 54 | 73 | 104 |
| 60 – 69 | 49 | 40 | 56 | 58 | 64 | 95 |
| 70 - 79 | 50 | 32 | 46 | 50 | 51 | 77 |
| <u>&gt;</u> 80 | 54 | 22 | 34 | 52 | 34 | 54 |

(Peters et al. 2011)

**Note:** The age category that applies for a subject at the Baseline visit will be used for the calculation of predicted grip values for all study time points.

#### **Walking Ability**

#### **Calculation of Predicted Six-Minute Walk Test Distance**

6MWT Distance (meters) = 868.8 - (2.99\*Age) - (74.7\*Gender)

Age in years. Men = 0 and Women = 1.

Gibbons WJ, Fruchter N, Sloan S, Levy RD. Reference Values for a Multiple Repetition 6-Minute Walk Test in Healthy Adults Older than 20 Years. J Cardpulm Rehabil. 2001 Mar/Apr; 21(2):87-93

**Note:** The age of a subject at the Baseline visit will be used for the calculation of 6MWT predicted values for all study time points.



Table 6: Regression Equations and Multiple Correlations of Sex, Age, and Weight with Muscle Strength (Newtons)

| Muscle Action | Side | Equation* | R | R <sup>2</sup> |
|---|---|---|---|---|
| Wrist extension | Non | 114.36 - 45.1S774A + .094W | .825 | .680 |
| | Dom | 123.65 - 48.5S784A + .092W | .826 | .683 |
| Elbow flexion | Non | 188.25 - 89.2\$650A + .132W | .882 | .779 |
| | Dom | 188.36 - 96.5S610A + .140W | .907 | .822 |
| Elbow extension | Non | 150.37 - 71.5S - 1.044A + .126W | .852 | .726 |
| | Dom | 156.49 - 73.0S - 1.032A + .116W | .853 | .727 |
| Shoulder lateral rotation | Non | 140.32 - 50.2S - 50.164A + .080W | .786 | .618 |
| | Dom | 147.66 - 54.5S930A + .088W | .810 | .656 |
| Shoulder extension | Non | 260.18 - 113.5S - 1.868A + .202W | .842 | .709 |
| | Dom | 278.99 - 120.0S - 1.99A + .202W | .855 | .731 |
| Shoulder abduction | Non | 165.16 - 74.9S910A + .126W | .843 | .710 |
| | Dom | 178.90 - 77.1S - 1.128A + .134W | .843 | .710 |
| Ankle dorsiflexion | Non | 302.54 - 60.9S - 2.203A + .159W | .742 | .550 |
| | Dom | 285.46 - 47.6S - 2.367A + .193W | .669 | .448 |
| Knee extension <sup>†</sup> | Non | 480.70 - 95.0S - 4.868A + .310W | .826 | .683 |
| | Dom | 465.22 - 84.7S - 4.803A + .325W | .820 | .673 |
| Hip flexion | Non | 216.48 - 74.6\$926A + .026W | .718 | .516 |
| • | Dom | 219.30 - 72.6S977A + .027W | .731 | .534 |
| Hip abdcution | Non | 203.32 - 73.3S - 1.247A + .192W | .794 | .630 |
| • | Dom | 195.24 - 62.4\$ - 1.184A + .198W | .764 | .584 |

<sup>\*</sup>S, sex (male = 0, female = 1); A, age (years); W, weight (Newtons).

Wrist extension (Bohannon 1997a)

<sup>&</sup>lt;sup>1</sup>The equations for knee extension are compromised by the upper limit of force (650N) recorded for 21 subjects.



# Pinch Strength Norms for Adults

# Average Performance of All Subjects on Key Pinch (kg.)

| | | | Men | | | Women | |
|-------|------|------|-----|----------|------|-------|----------|
| Age | Hand | Mean | SD | Range | Mean | SD | Range |
| 20-24 | R | 11.8 | 1.6 | 9.5-15.4 | 8.0 | 0.9 | 6.4-10.4 |
| | L | 11.2 | 1.5 | 8.6-14.1 | 7.3 | 1.0 | 5.9-10.4 |
| 25-29 | R | 12.1 | 2.2 | 8.6-18.6 | 8.0 | 1.0 | 6.4-10.0 |
| | L | 11.3 | 2.0 | 8.6-17.7 | 7.5 | 1.0 | 5.9-10.0 |
| 30-34 | R | 12.0 | 2.2 | 9.1-16.3 | 8.5 | 1.4 | 5.9-11.3 |
| | L | 11.9 | 2.3 | 7.7-16.3 | 8.1 | 1.6 | 5.4-11.8 |
| 35-39 | R | 11.8 | 1.5 | 9.5-14.5 | 7.5 | 0.9 | 5.4-9.5 |
| | L | 11.6 | 1.8 | 8.2-14.5 | 7.3 | 1.2 | 5.4-10.0 |
| 40-44 | R | 11.6 | 1.2 | 9.5-14.1 | 7.6 | 1.4 | 4.5-10.9 |
| | L | 11.4 | 1.8 | 8.6-14.1 | 7.2 | 1.4 | 3.6-10.0 |
| 45-49 | R | 11.7 | 1.8 | 8.6-15.9 | 8.0 | 1.5 | 5.9-10.9 |
| | L | 11.2 | 2.0 | 8.2-19.1 | 7.5 | 1.3 | 5.4-10.9 |
| 50-54 | R | 12.1 | 2.0 | 9.1-15.4 | 7.6 | 1.1 | 5.4-10.0 |
| | L | 11.8 | 1.9 | 9.1-16.8 | 7.3 | 1.2 | 5.4-10.0 |
| 55-59 | R | 11.0 | 1.9 | 8.2-15.4 | 7.1 | 1.1 | 5.0-9.5 |
| | L | 10.4 | 2.1 | 5.9-14.1 | 6.7 | 1.0 | 5.4-8.6 |
| 60-64 | R | 10.5 | 2.4 | 6.4-16.8 | 7.0 | 1.2 | 4.5-9.1 |
| | L | 10.1 | 1.9 | 7.3-15.0 | 6.4 | 1.1 | 4.5-8.6 |
| 65-69 | R | 10.6 | 1.8 | 7.7-14.5 | 6.8 | 1.2 | 4.5-9.5 |
| | L | 10.0 | 1.6 | 7.7-12.7 | 6.5 | 1.3 | 4.5-9.1 |
| 70-74 | R | 8.8 | 1.1 | 7.3-11.3 | 6.6 | 1.3 | 3.6-10.0 |
| | L | 8.7 | 1.4 | 5.9-12.7 | 6.3 | 1.4 | 4.1-10.0 |
| 75 + | R | 9.3 | 2.1 | 4.1-14.1 | 5.7 | 1.0 | 3.6-7.7 |
| | L | 8.7 | 1.4 | 5.9-10.9 | 5.2 | 1.2 | 3.2-7.3 |

The above information is taken from <u>Grip & Pinch Strength: Normative Data</u> <u>for Adults</u>, Arch Phys Med Rehabil 66:69-72, 1985, V. Mathiowetz,et al



# 10.4 Summary of Efficacy Assessment in Parent Studies and in Current Study CL302

| Study | Functional Test | Questionnaire | Biomarker |
|---|---|---|---|
| CL-202 | Week 0, 12, 36, 60, 84, 108, 132, 156 | Week 0, 12, 36, 84, 156 | Week 0, 12, 16, 36, 60, 108, 156 |
| | Muscle strength as measured by HHD; Walking ability as measured by the 6MWT; Arm raising ability as measured by the weighted arm lift test; Functional disability as measured by the GNEM-FAS. | None | CK Free Serum SA Free and total urine SA (Part I only, Week 0, 12) Serum protein markers (Part I only, Week 0, 12) |
| CL-301 | Week 8, 16, 24, 32, 40, 48 | Week 8, 16, 24, 32, 40, 48 | Week0, 8, 16, 24, 32, 40, 48 |
| | Muscle strength as measured by HHD; Walking ability as measured by the 6MWT; Arm raising ability as measured by the weighted arm lift test; Muscle strength on mobility domain score by GNEM-FAS | The total score on a 45-item self-report of INQoL. Week 24, 48 The CGI Severity scale (CGI-S, baseline only), and improvement scale (CGI-I, at each subsequent visit). | CK Serum SA Week0, 16, 32, 48 Free, total and bound urine SA Urine ManNAc |
| CL-203 | Week 0, 12, 24, 36, 48 | Week 0, 12, 24, 36, 48 | Week 0, 12, 24, 36, 48 |
| | Muscle strength by GNEM-FAS Expanded Version total score; Upper extremity strength as measured by HHD Lower extremity muscle strength as measured by HHD | Health-related quality of life as assessed by SF-36 Symptom severity as measured by PGI-S (baseline only) and PGI-C (at each subsequent visit) | CK Free serum SA Serum aceneuramic acid Free, total and bound Urine SA Urine ManNAc |
| CL-302 | Week 0, 8, 16, 24, 48, 72, 96 | Week 0, 8, 16, 24, 48, 72, | Week 0, 8, 16, 24, 48, 72, 96 |
| (Patients<br>from<br>202/301) | Muscle strength as measured by HD; Walking ability as measured by the 6MWT; Arm raising ability as measured by the weighted arm lift test; Change in muscle strength on mobility domain score by | The total score on a 45-item self-report of INQoL. | CK Free serum SA. Urine ManNAc |



| Study | Functional Test | Questionnaire | Biomarker |
|---|---|---|---|
| CL-302 | Week 0, 24, 48, 72, 96 | Week 0, 24, 48, 72, 96 | Week 0, 8, 16, 24, 48, 72, 96 |
| (Patients from CL203) | Muscle strength in GNEM-FAS<br>Expanded Version total score;<br>Muscle strength as measured by<br>HHD. | Health-related quality of life as assessed by SF-36 | CK Free serum SA. Urine ManNAc |



# 10.5 Schedule of Events

| ASSESSMENTS AND EVENTS* | SCREENING/<br>BASELINE <sup>a</sup> | TREATMENT PERIOD | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | MONTH 2<br>(WEEK 8)<br>VISIT<br>(± 5 DAYS)‡ | MONTH 4<br>(WEEK 16)<br>VISIT<br>(± 5 DAYS) ‡ | MONTH 6<br>(WEEK 24)<br>VISIT<br>(± 5 DAYS) | MONTH 12 VISIT (WEEK 48) (± 2WEEKS) | MONTH 18<br>VISIT<br>(WEEK 72)<br>(± 2WEEKS) | MONTH 24 (WEEK 96) OR EARLY TERMINATION VISIT (± 2WEEKS) | SAFETY<br>FOLLOW<br>UP (+ 5<br>DAYS) <sup>m</sup> |
| SAFETY ASSESSMENTS (ALL SUBJECTS) | | | | | | | | |
| INFORMED CONSENT | X | | | | | | | |
| MEDICAL HISTORY | X | | | | | | | |
| INTERVAL HISTORY b | X | X | X | X | X | X | X | |
| PHYSICAL EXAMINATION <sup>c</sup> | X | X | X | X | X | X | X | |
| VITAL SIGNS | X | X | X | X | X | X | X | |
| HEMATOLOGY, CHEMISTRY PANEL,<br>URINALYSIS | X | X | X | X | X | X | X | |
| PREGNANCY TEST | X | X | X | X | X | X | X | |
| CONCOMITANT MEDICATIONS | X | X | X | X | X | X | X | X |
| SUICIDAL IDEATION AND BEHAVIOR (C-SSRS) d | X | X | X | X | X | X | X | |
| Adverse events | X | X | X | X | X | X | X | X |
| PHARMACODYNAMIC ASSESSMENTS (ALL S | UBJECTS) | | | | | | | |
| BIOMARKERS: CK, FREE SERUM SA, AND<br>BIOMARKERS OF SIALYATION AND OTHER<br>BIOMARKERS <sup>c</sup> | X | X | X | X | X | X | X | |
| FREE, TOTAL AND BOUND URINE SA LEVELS <sup>f</sup> | X | X | X | X | X | X | X | |
| URINE TEST FOR MANNAC <sup>g</sup> | X | X | X | X | X | X | X | |

Proprietary and Confidential Page 39



| ASSESSMENTS AND EVENTS* | SCREENING/<br>BASELINE <sup>a</sup> | TREATMENT PERIOD | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | MONTH 2<br>(WEEK 8)<br>VISIT<br>(± 5 DAYS)‡ | MONTH 4<br>(WEEK 16)<br>VISIT<br>(± 5 DAYS) ‡ | MONTH 6<br>(WEEK 24)<br>VISIT<br>(± 5 DAYS) | MONTH 12<br>VISIT (WEEK<br>48)<br>(± 2WEEKS) | MONTH 18<br>VISIT<br>(WEEK 72)<br>(± 2WEEKS) | MONTH 24 (WEEK 96) OR EARLY TERMINATION VISIT (± 2WEEKS) | SAFETY<br>FOLLOW<br>UP (+ 5<br>DAYS) <sup>m</sup> |
| TREATMENT DISPENSING AND COMPLIANCE | E (ALL SUBJEC | CTS) | | | | | | |
| TREATMENT DISPENSED h | X | X | X | X | X | X | | |
| TREATMENT COMPLIANCE | | X | X | X | X | X | X | |
| EFFICACY ASSESSMENTS (UX001-CL202 AND ADDRESS OF THE PROPERTY | ND UX001-CL | 301 SUBJECTS | s) <sup>i</sup> | | | | | |
| DYNAMOMETRY | X | X | X | X | X | X | X | |
| 6-MINUTE WALK TEST (6MWT) | X | X | X | X | X | X | X | |
| SIT-TO-STAND TEST | X | X | X | X | X | X | X | |
| WEIGHTED ARM LIFT TEST | X | X | X | X | X | X | X | |
| GNE MYOPATHY FUNCTIONAL<br>ACTIVITIES SCALE (GNEM-FAS) | X | X | X | X | X | X | X | |
| INDIVIDUALIZED NEUROMUSCULAR<br>QUALITY OF LIFE QUESTIONNAIRE<br>(INQOL) | X | X | X | X | X | X | X | |
| EFFICACY ASSESSMENTS (UX001-CL203 St | UBJECTS) | | | | | | | |
| Dynamometry <sup>j</sup> | X | | | X | X | X | X | |
| GNEM-FAS k | X | | | X | X | X | X | |
| SHORT FORM HEALTH SURVEY-36 (SF-36) | X | | | X | X | X | X | |

Refer to study-related materials for recommended timing and order of assessments to be administered at each study visit.

<sup>\$\</sup>frac{1}{2}\$ Subjects who roll-over from the UX001-CL203 study will not have a Month 2 or Month 4 visit. Assessments at these visits will only be performed for subjects who roll-over from the UX001-CL202 and UX001-CL301 studies. UX001-CL202 subjects will complete the same efficacy assessments as the subjects who rollover from UX001-CL301.



- a. Potential subjects can be screened up to 5 days after the last dose on the parent study. Baseline Visit should be not be more than 5 days after Screening visit. Subjects can have a concurrent Screening and Baseline visits. Study drug will be dispensed only after all study procedures at the Baseline Visit have been performed. For subjects who discontinue prior to completing the study, every reasonable effort should be made to perform the Early Termination (ET) procedures within four weeks of discontinuation.
- b. Interval history will include any signs, symptoms, or events (i.e. falls) experienced by the subject since the prior study visit that are not related to study procedure(s) performed at prior study visits or study drug. Interval history may include exacerbation or improvement in existing medical conditions (including the clinical manifestations of GNEM) that might interfere with study participation, safety, and/or positively or negatively impact performance of functional assessments.
- c. The physical examinations at Baseline/Screening, including a neurological examination; all others will be brief physical examinations. If a patient is unable to stand or has significant postural issues that interfere with collection of a standing height, self-reported adult height should be captured.
- d. Baseline C-SSRS administered at Baseline/Screening visit (may be same as last visit in parent study). Since Last Visit C-SSRS administered at all subsequent visits.
- e. Serum will be obtained at all study visits to evaluate creatine kinase (CK), serum SA and potential biomarkers of sialylation, and other markers of muscle injury and remodeling.
- f. Blood samples, preferably pre dose, and first-morning void urine will be collected to assess trough SA levels; record volume of urine collected.
- g. An aliquot from first morning void urine will be used for assessment of ManNAc; record volume of urine collected.
- h. Subjects should be instructed to return unused study drug and packaging to every visit. Note that all subjects being treated with 12 g/day Ace-ER in UX001-CL202 will be transitioned to 6 g/day Ace-ER dose in this protocol.
- i. For UX001-CL202 subjects, assessments that cannot be safely performed by a subject due to disease progression should not be administered.
- j. For subjects enrolling from UX001-CL203, lower extremity muscle strength for knee extensors muscle group only.
- k. For subjects enrolling from UX001-CL203, the GNEM-FAS Expanded version will be used.
- l. The Early Termination Visit occurs if a subject discontinues prior to completing the study or no longer wants to participate in the study. Every reasonable effort should be made to have subjects return to the clinic within 4 weeks of discontinuation and perform the Early Termination procedures; however, subjects who are unable to return to the clinic will be given the option of having an Early Termination Visit telephone call within 4 weeks of discontinuation from study, where appropriate information will be collected by the clinical site.
- m. Safety Follow-up visit to be conducted by phone 30 days (+5 days) after last dose of study drug.



# 10.6 Adverse Events to Monitor

# 10.6.1 Gastrointestinal MedDRA Query

The following MedDRA PTs are included in the gastrointestinal SMQ version 17.1.

| Narrow Scope | Broad Scope |
|----------------------------------|--------------------------------------|
| Abdominal discomfort | Anorectal swelling |
| Abdominal distension | Antacid therapy |
| Abdominal pain | Antidiarrhoeal supportive care |
| Abdominal pain lower | Antiemetic supportive care |
| Abdominal pain upper | Breath odour |
| Abdominal symptom | Chest pain |
| Abdominal tenderness | Colonic lavage |
| Abnormal faeces | Dysphagia |
| Aerophagia | Early satiety |
| Anorectal discomfort | Gastritis prophylaxis |
| Bowel movement irregularity | Gastrointestinal disorder therapy |
| Change of bowel habit | Gastrointestinal tract irritation |
| Constipation | Gastrooesophageal reflux prophylaxis |
| Defaecation urgency | Glycogenic acanthosis |
| Diarrhoea | Hypovolaemia |
| Epigastric discomfort | Laxative supportive care |
| Eructation | Malabsorption |
| Faecal volume decreased | Mucous stools |
| Faecal volume increased | Oesophageal polymer implantation |
| Faeces hard | Pernicious anaemia |
| Faeces soft | Post procedural constipation |
| Flatulence | Post procedural diarrhea |
| Frequent bowel movements | Post-tussive vomiting |
| Gastrointestinal pain | Probiotic therapy |
| Gastrointestinal sounds abnormal | Procedural nausea |
| Gastrointestinal toxicity | Procedural vomiting |
| Infrequent bowel movements | Prophylaxis against diarrhoea |
| Nausea | Prophylaxis of nausea and vomiting |
| Non-cardiac chest pain | Regurgitation |
| Oesophageal discomfort | Retching |
| Oesophageal pain | Steatorrhoea |
| Premenstrual cramps | Vomiting projectile |
| Vomiting | |



# 10.6.2 Liver-Related Investigations

The following MedDRA PTs are included in the category "liver-related investigations."

Alanine aminotransferase abnormal

Alanine aminotransferase increased

Aspartate aminotransferase abnormal

Aspartate aminotransferase increased

Gamma-glutamyl transferase abnormal

Gamma-glutamyl transferase increased

Hepatic enzyme abnormal

Hepatic enzyme increased

Liver function test abnormal

Transaminases abnormal

Transaminases increased



# 10.7 Table templates for efficacy and safety analysis presentation

Table 14.x.x.x

Summary of HHD Upper Extremity Component (UEC) Scores - Parent Study CL301

(Full Analysis Set)

| | ACE-ER 6 g/day | | | | |
|---|---|---|---|---|---|
| | Treatment in Pa | arent Study CL301 | Treat | ment in Parent Stud | dy CL301 |
| | (Parent stu | ıdy baseline) | ( | Current study basel | ine) |
| Visit | Placebo | Ace-ER 6 g/day | Placebo | Ace-ER 6 g/day | Total |
| Statistics | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| Week 8 | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | xx.xxx | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| Median | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Change from Baseline to Week 8 | | | | | |
| <b></b> | | | | | |
| Week 96 | | | | | |

SD=standard deviation.

Study UX001-CL301 is a placebo-controlled efficacy study.



# Table 14.x.x.x Summary of HHD Upper Extremity Component (UEC) Scores - Parent Study CL202 (Full Analysis Set)

| | Ace-ER 6 g/day |
|--------------------------------|------------------------|
| Visit | Current Study Baseline |
| Statistics | (N=xx) |
| eek 8 | |
| n | xx |
| Mean | XX.XX |
| SD | xx.xxx |
| Median | xx.xx |
| Min, Max | xx.x, xx.x |
| Change from Baseline to Week 8 | |
| eek 96 | |

SD=standard deviation.

Study UX001-CL202 is an extension study of CL201 with 10 naïve subjects.



# Table 14.x.x.x Summary of HHD Individual Raw Strength Scores: Knee Extensors - Parent Study CL203 (Full Analysis Set)

| | Ace-ER 6 g/day | |
|---|---|---|
| /isit | Parent Study Baseline | Current Study Baseline |
| Statistics | (N=xx) | (N=xx) |
| Jeek 24 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX,XXX | XX.XXX |
| Median | XX.XX | XX.XX |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline to Week 24 | | |
| <br>leek 96 | | |

SD=standard deviation, Min=minimum, Max=maximum. Study UX001-CL203 is a safety study.



# Table 14.x.x.x Overall Summary of Treatment Emergent Adverse Events (Safety Analysis Set)

| | Ace-ER 6 g/day | | | | | |
|---|---|---|---|---|---|---|
| _ | Treatment in Parent Study CL301 Parent Study | | | | | |
| _ | | Ace-ER 6 | | | | Total |
| | Placebo | g/day | All | CL202 | CL203 | (N=xx) |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | |
| Number of subjects with TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum severity | | | | | | |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of subjects with treatment-<br>related TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of serious TEAEs | XX | xx | XX | XX | XX | xx |
| Number of subjects with serious<br>TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of TEAEs causing<br>discontinuation | xx | XX | xx | XX | xx | XX |
| Number of subjects with TEAEs causing discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |